CLINICAL TRIAL: NCT05723302
Title: The Effect of Resistant Proprioceptive Neuromuscular Facilitation Exercises on Respiratory Muscle Strength in Chronic Obstructive Pulmonary Diseases
Brief Title: Chronic Obstructive Pulmonary Diseases and Proprioceptive Neuromuscular Facilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Mehmet Akif Ersoy Canakkale State Hospital (Other Government); Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, sevda vurur, Student, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulMUH_1999
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal Inspiratory Pressure (Experimental): MIP Maximal Inspiratory Pressure
  Interventions: Diagnostic Test: MIP/MEP
- Maximal Expiratory Pressure (Experimental): MEP Maximal Expiratory Pressure
  Interventions: Diagnostic Test: MIP/MEP

INTERVENTIONS:
Diagnostic Test: MIP/MEP — MIP/MEP

SUMMARY:
To investigate the effects of resistant proprioceptive neuromuscular facilitation exercises on physical fitness, respiratory muscle strength, walking distance and quality of life in chronic obstructive pulmonary patients.

DETAILED DESCRIPTION:
The study was carried out between January 2017 and January 2019, with patients followed up with the diagnosis of COPD in Çanakkale Mehmet Akif Ersoy State Hospital and Çanakkale Onsekiz Mart University Medical Faculty Hospital, Department of Chest Diseases. It was approved by Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee (Date: 30.12.2016, Decision No. 573) and was done in accordance with the Declaration of Helsinki. All participants were informed about the purpose of the study, the total duration of treatment and the applications to be made, and a consent form was signed. The study was conducted as a prospective and randomized controlled study, and inclusion and exclusion criteria were determined.

Thirty-five patients diagnosed with COPD were referred to the study, four patients were excluded because they did not meet the inclusion criteria, and the study was conducted with a total of 31 participants.

The 31 patients included in the study were randomized after their initial evaluation and divided into two groups as experimental and control groups. Patients meeting the inclusion criteria were divided into 2 groups. Randomized by ordering by date of application.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with stage 1, stage 2 and stage 3 COPD according to GOLD (Global Initiative for Obstructive Lung Diseases) criteria
* Having FEV1/FVC <70% according to pulmonary function test
* Being clinically stable
* Being over 18 years old
* Volunteer to participate in the program

Exclusion Criteria:

* Having a COPD exacerbation in the last 8 weeks
* To have participated in a regular exercise training program in the last 1 year
* Having a musculoskeletal disease and neuromuscular disease that may prevent exercise
* Inability to cooperate for pulmonary function test and respiratory muscle strength measurement
* Being on long-term oxygen therapy

Ages: 38 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
HADS | 10 minutes
  Hospital Anxiety Depression Scale

SECONDARY OUTCOMES:
SGRQ | 15 minutes
  St George's Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mehmet Akif Ersoy State Hospital, Çanakkale
  - Çanakkale Onsekiz Mart University, Çanakkale

IPD SHARING:
Plan to Share IPD: No